CLINICAL TRIAL: NCT03809182
Title: Effect of Dexmedetomidine on Postoperative Glucose Levels and Insulin Secretion Patterns in Obese Patients With Impaired Glucose Tolerance.
Brief Title: Effect of Dexmedetomidine on Postoperative Glucose and Insulin Levels.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, Eduardo Vega, Instructor, Pontificia Universidad Catolica de Chile
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Dexmedetomidine and glycemia.
Record Dates: First submitted 2018-12-30; First posted 2019-01-18 (Actual); Results first posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Bariatric Surgery Candidate; Glucose Intolerance; Insulin Resistance
Keywords: Impaired Glucose Tolerance; Obese patients; Dexmedetomidine
MeSH Terms: conditions — Glucose Intolerance; Insulin Resistance | interventions — Dexmedetomidine; Sodium Chloride; Saline Solution; Fentanyl; Morphine

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (2):
- Dexmedetomidine (Experimental): After anesthesia induction, patients who were randomized to the Dexmedetomidine group received a bolus of 1ug/kg in 10 minutes, followed by an infusion of 0.5ug/kg/h until the end of surgery. In the case of intraoperative increment of the blood pressure and/or heart rate more than 25% from its baseline, fentanyl 1ug/kg was administered.
  Interventions: Drug: Dexmedetomidine; Drug: Fentanyl; Drug: Morphine Sulfate
- 0.9% Sodium-chloride (Placebo Comparator): After anesthesia induction, patients who were randomized to the Placebo group received a bolus and infusion of 0.9% normal saline at the same rate as the Dexmedetomidine group until the end of surgery. In the case of intraoperative increment of the blood pressure and/or heart rate more than 25% from its baseline, fentanyl 1ug/kg was administered.
  Interventions: Drug: 0.9% Sodium-chloride; Drug: Fentanyl; Drug: Morphine Sulfate

INTERVENTIONS:
Drug: Dexmedetomidine — A bolus of 1ug/kg in 10 minutes, followed by an infusion of 0.5ug/kg/h until the end of surgery.
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: 0.9% Sodium-chloride — The same infusion rate used in the dexmedetomidine group.
  Other Names: Normal saline
  Arms: 0.9% Sodium-chloride
Drug: Fentanyl — Intraoperative fentanyl was given in case of 25% increment in the blood pressure and/or heart rate in comparison to baseline (previous anesthesia induction).
  Other Names: Sublimaze
Drug: Morphine Sulfate — Boluses of 3mg of intravenous morphine were given in the postoperative acute care unit. Once the pain score was equal or less than 3/10 the patient-controlled analgesia pumps were installed and the patients were discharged to their room.
  Other Names: Morphine

SUMMARY:
This study investigated the effect of dexmedetomidine in obese patients undergoing bariatric surgery.

DETAILED DESCRIPTION:
A prospective, double-blind, randomized controlled trial was performed. Consenting obese adult patients with impaired glucose tolerance, undergoing bariatric surgery, were randomized, by a computer, to receive placebo (0.9% Sodium-chloride) or dexmedetomidine 1 ug/kg bolus in 10 minutes followed by an infusion of 0.5 ug/kg/h until the end of surgery. Baseline HgbA1c, glucose, and insulin plasmatic levels were measured. Subsequently, glucose and insulin levels were taken every 2 hours during the first 12 hours from the onset of the drug infusion. Intraoperative fentanyl and postoperative morphine consumption, pain score, the occurrence of emesis, and postoperative sedation levels were recorded as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Obese patient (BMI>30)
* American Society of Anesthesiologists grades II or III
* Diagnosis of impaired glucose tolerance
* Undergoing sleeve gastrectomy

Exclusion Criteria:

* Baseline glucose > 200mg/dl
* Diagnosis of Diabetes
* Under corticosteroids treatment
* Oral hypoglycemic medication within 7 days previous surgery
* Use of insulin within 24h previous surgery
* Allergy to any drug used in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-09-27 (Actual); Primary Completion 2013-07-25 (Actual); Study Completion 2013-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio Ibacache, MD, PhD, Study Director — Pontificia Universidad Catolica de Chile

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patients were recruited at the Pontifical Catholic University Hospital between 2012 and 2013. Twenty patients were assigned to each arm to allow some dropouts. Nonetheless, every randomized patient included in the study was analyzed at the end of it (intention to treat analysis).
Pre-assignment Details: No patient was excluded from the study after being assigned to one arm/group.
Groups:
- Dexmedetomidine: After anesthesia induction, patients who were randomized to the Dexmedetomidine group received:
  Dexmedetomidine: A bolus of 1ug/kg in 10 minutes, followed by an infusion of 0.5ug/kg/h until the end of surgery.
  Fentanyl: Intraoperative fentanyl was given in case of 25% increment in the blood pressure and/or heart rate in comparison to baseline (previous anesthesia induction).
  Morphine Sulfate: Boluses of 3mg of intravenous morphine were given in the postoperative acute care unit. Once the pain score was equal or less than 3/10 the patient-controlled analgesia pumps were installed and the patients were discharged to their room.
- 0.9% Sodium-chloride: After anesthesia induction, patients who were randomized to the Placebo group received:
  0.9% Sodium-chloride: The same bolus and infusion rate used in the dexmedetomidine group.
  Fentanyl: Intraoperative fentanyl was given in case of 25% increment in the blood pressure and/or heart rate in comparison to baseline (previous anesthesia induction).
  Morphine Sulfate: Boluses of 3mg of intravenous morphine were given in the postoperative acute care unit. Once the pain score was equal or less than 3/10 the patient-controlled analgesia pumps were installed and the patients were discharged to their room.
Period: Overall Study
Arm/Group | Dexmedetomidine | 0.9% Sodium-chloride
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics from the entire study population were measured.
Groups:
- Dexmedetomidine: After anesthesia induction, patients who were randomized to the Dexmedetomidine group, received a bolus of 1ug/kg in 10 minutes, followed by an infusion of 0.5ug/kg/h until the end of surgery. In the case of intraoperative increment of the blood pressure and/or heart rate more than 25% from its baseline, fentanyl 1ug/kg was administered.
  Dexmedetomidine: A bolus of 1ug/kg in 10 minutes, followed by an infusion of 0.5ug/kg/h until the end of surgery.
  Fentanyl: Intraoperative fentanyl was given in the case of 25% increment in the blood pressure and/or heart rate in comparison to baseline (previous anesthesia induction).
  Morphine Sulfate: Boluses of 3mg of intravenous morphine were given in the postoperative acute care unit. Once the pain score was equal or less than 3/10 a patient-controlled analgesia pump was installed and the patient was discharged to his/her room.
- 0.9% Sodium-chloride: After anesthesia induction, patients who were randomized to the Placebo group received a bolus and infusion of 0.9% normal saline at the same rate as the Dexmedetomidine group until the end of surgery. In the case of intraoperative increment of the blood pressure and/or heart rate more than 25% from its baseline, fentanyl 1ug/kg was administered.
  0.9% Sodium-chloride: The same dose used in the dexmedetomidine group (bolus and infusion).
  Fentanyl: Intraoperative fentanyl was given in the case of 25% increment in the blood pressure and/or heart rate in comparison to baseline (previous anesthesia induction).
  Morphine Sulfate: Boluses of 3mg of intravenous morphine were given in the postoperative acute care unit. Once the pain score was equal or less than 3/10 a patient-controlled analgesia pump was installed and the patient was discharged to his/her room.
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine | 0.9% Sodium-chloride | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (10.2) | 31.5 (9.9) | 32 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 15 | 35
  Male | 0 | 5 | 5
Region of Enrollment [Number; unit: participants]
  Chile | 20 | 20 | 40
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 34.4 (2.5) | 35.2 (3.6) | 34.8 (3.1)
ASA physical status II [Count of Participants; unit: Participants] — ASA I A normal healthy patient, ASA II A patient with mild systemic disease, ASA III A patient with severe systemic disease, ASA IV A patient with severe systemic disease that is a constant threat to life, ASA V A moribund patient who is not expected to survive without the operation, ASA VI A declared brain-dead patient whose organs are being removed for donor purposes
  Participants | 20 | 20 | 40
Risk score for postoperative nausea and vomiting (PONV) in adults [Count of Participants; unit: Participants] — This corresponds to the Apfel simplified risk score, which is based on 4 predictors: female sex, history of PONV and/or motion sickness, nonsmoking status, and use of postoperative opioids. The higher the number of risk factors the more probable the incidence of PONV.
  Participants
    0 risk factor | 0 | 0 | 0
    1 risk factor | 0 | 4 | 4
    2 risk factors | 14 | 9 | 23
    3 risk factors | 5 | 6 | 11
    4 risk factors | 1 | 1 | 2
Baseline HbA1c [Mean (Standard Deviation); unit: Percentage] | 5.4 (0.2) | 5.4 (0.4) | 5.4 (0.3)

OUTCOME MEASURES:

1. Primary Outcome: Plasmatic Glucose Levels (mg/dl).
Description: Change of baseline glucose levels within the first 12 postoperative hours.
Time Frame: Baseline levels(T0) and at hour 2(T1), 4(T2), 6(T3), 8(T4), 10(T5), and 12(T6) after the onset of bolus and infusion of dexmedetomidine
Population: All recruited population was analyzed.
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- 0.9% Sodium-chloride: After anesthesia induction, patients who were randomized to the Placebo group received:
  0.9% Sodium-chloride: The same rate infusion used in the dexmedetomidine group (bolus and infusion).
  Fentanyl: Intraoperative fentanyl was given in case of 25% increment in the blood pressure and/or heart rate in comparison to baseline (previous anesthesia induction).
  Morphine Sulfate: Boluses of 3mg of intravenous morphine were given in the postoperative acute care unit. Once the pain score was equal or less than 3/10 a patient-controlled analgesia pumps were installed and the patients were discharged to their room.
Arm/Group | Dexmedetomidine | 0.9% Sodium-chloride
Number analyzed (Participants) | 20 | 20
mg/dl
  Baseline level (T0) | 80 (15) | 82 (8)
  Hour 2 (T1) | 114 (29) | 111 (20)
  Hour 4 (T2) | 124 (25) | 129 (17)
  Hour 6 (T3) | 131 (60) | 120 (16)
  Hour 8 (T4) | 122 (41) | 118 (17)
  Hour 10 (T5) | 130 (62) | 117 (18)
  Hour 12 (T6) | 125 (31) | 117 (17)
Statistical Analysis 1: Comparison: Dexmedetomidine vs 0.9% Sodium-chloride; Null hypothesis: There is no difference in plasmatic glucose levels between dexmedetomidine and 0.9% sodium-chloride groups; Test type: Superiority; p = 0.38, Mixed Models Analysis — A p-value less than .05 was considered statistically significant

2. Primary Outcome: Plasmatic Insulin Levels (uU/ml).
Description: Change of baseline insulin levels within the first 12 postoperative hours.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: uU/dl
Groups:
- Dexmedetomidine: After anesthesia induction, patients who were randomized to the Dexmedetomidine group, received a bolus of 1ug/kg in 10 minutes, followed by an infusion of 0.5ug/kg/h until the end of surgery. In case of intraoperative increment of the blood pressure and/or heart rate more than 25% from its baseline, fentanyl 1ug/kg was administered.
  Dexmedetomidine: A bolus of 1ug/kg in 10 minutes, followed by an infusion of 0.5ug/kg/h until the end of surgery.
  Fentanyl: Intraoperative fentanyl was given in case of 25% increment in the blood pressure and/or heart rate in comparison to baseline (previous anesthesia induction).
  Morphine Sulfate: Boluses of 3mg of intravenous morphine were given in the postoperative acute care unit. Once the pain score was equal or less than 3/10 a patient-controlled analgesia pumps were installed and the patients were discharged to their room.
- 0.9% Sodium-chloride: After anesthesia induction, patients who were randomized to the Placebo group received a bolus and infusion of 0.9% normal saline at the same rate as the Dexmedetomidine group until the end of surgery. In case of intraoperative increment of the blood pressure and/or heart rate more than 25% from its baseline, fentanyl 1ug/kg was administered.
  0.9% Sodium-chloride: The same dose used in the dexmedetomidine group (bolus and infusion).
  Fentanyl: Intraoperative fentanyl was given in case of 25% increment in the blood pressure and/or heart rate in comparison to baseline (previous anesthesia induction).
  Morphine Sulfate: Boluses of 3mg of intravenous morphine were given in the postoperative acute care unit. Once the pain score was equal or less than 3/10 a patient-controlled analgesia pumps were installed and the patients were discharged to their room.
Arm/Group | Dexmedetomidine | 0.9% Sodium-chloride
Number analyzed (Participants) | 20 | 20
uU/dl
  Baseline level (T0) | 10.5 (6) | 11.2 (6)
  Hour 2 (T1) | 11.8 (9) | 19.9 (11.8)
  Hour 4 (T2) | 16.7 (9.5) | 30.3 (19.9)
  Hour 6 (T3) | 16.8 (11.4) | 23 (11.4)
  Hour 8 (T4) | 16.6 (8.9) | 21.5 (10.4)
  Hour 10 (T5) | 16 (10) | 24 (17.7)
  Hour 12 (T6) | 16.6 (9.2) | 25.9 (18.3)
Statistical Analysis 1: Comparison: Dexmedetomidine vs 0.9% Sodium-chloride; Null hypothesis: There is no difference in insulin levels between dexmedetomidine and 0.9% sodium-chloride groups; Test type: Superiority; p = 0.02, Mixed Models Analysis — A p-value less than .05 was considered statistically significant

3. Secondary Outcome: Fentanyl Consumption.
Description: Amount of fentanyl (ug/kg) intraoperatively administered.
Time Frame: Since the beginning of anesthesia until the end of it, an average of one hour and a half.
Measure: Mean (Standard Deviation); unit: mcg/kg
Arm/Group | Dexmedetomidine | 0.9% Sodium-chloride
Number analyzed (Participants) | 20 | 20
mcg/kg | 6.0 (2.2) | 7 (2.4)

4. Secondary Outcome: Amount (mg) of Morphine Consumed.
Description: Morphine consumption in the first 24 postoperative hours.
Time Frame: At 24h postoperative hours.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Dexmedetomidine | 0.9% Sodium-chloride
Number analyzed (Participants) | 20 | 20
mg | 26 (14.4) | 18.4 (10.6)

5. Secondary Outcome: Pain Scores in the First 24 Postoperative Hours.
Description: Visual analogue scale (VAS), provided by patients, ranging from 0 to 10 (0= no pain and 10= worst possible pain). We considered a pain score between 1-3, 4-6 and 7-10 as mild, moderate and severe pain, respectively.
Time Frame: At postoperative hours 2(T1), 4(T2), 6(T3), 8(T4), 10(T5), 12(T6) and 24(T7).
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Dexmedetomidine | 0.9% Sodium-chloride
Number analyzed (Participants) | 20 | 20
units on a scale
  Hour 2 (T1) Pain at rest | 0 [0 to 2] | 0 [0 to 4]
  Hour 2 (T1) Pain at movement | 0 [0 to 2] | 0 [0 to 5]
  Hour 4 (T2) Pain at rest | 4 [2 to 5] | 3 [2 to 4]
  Hour 4 (T2) Pain at movement | 5 [4 to 6] | 4 [3 to 6]
  Hour 6 (T3) Pain at rest | 3 [1 to 5] | 2 [2 to 3]
  Hour 6 (T3) Pain at movement | 4 [2 to 6] | 4 [2 to 5]
  Hour 8 (T4) Pain at rest | 3 [1 to 5] | 1 [0 to 3]
  Hour 8 (T4) Pain at movement | 4 [3 to 7] | 4 [2 to 4]
  Hour 10 (T5) Pain at rest | 3 [1 to 4] | 1 [0 to 2]
  Hour 10 (T5) Pain at movement | 5 [3 to 6] | 3 [2 to 5]
  Hour 12 (T6) Pain at rest | 3 [0 to 4] | 1 [0 to 2]
  Hour 12 (T6) Pain at movement | 3 [2 to 5] | 3 [2 to 4]
  Hour 24 (T7) Pain at rest | 2 [0 to 3] | 0 [0 to 2]
  Hour 24 (T7) Pain at movement | 3 [1 to 4] | 3 [1 to 3]

6. Secondary Outcome: Sedation-agitation Scores in the First 12 Postoperative Hours.
Description: Sedation-agitation scale (SAS), ranging from 1 to 7 (1=unarousable, 2=very sedated, 3=sedated, 4=calm and cooperative, 5=agitated, 6=very agitated and 7=dangerous agitation).
Time Frame: At postoperative hours 2(T1), 4(T2), 6(T3), 8(T4), 10(T5) and 12(T6).
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Dexmedetomidine | 0.9% Sodium-chloride
Number analyzed (Participants) | 20 | 20
score on a scale
  Hour 2 (T1) | 3 [3 to 4] | 4 [4 to 4]
  Hour 4 (T2) | 4 [3 to 4] | 4 [4 to 4]
  Hour 6 (T3) | 4 [4 to 4] | 4 [4 to 4]
  Hour 8 (T4) | 4 [4 to 4] | 4 [4 to 4]
  Hour 10 (T5) | 4 [4 to 4] | 4 [4 to 4]
  Hour 12 (T6) | 4 [4 to 4] | 4 [4 to 4]

7. Secondary Outcome: Postoperative Nausea and Vomiting.
Description: Number of patients with postoperative nausea and vomiting in the first 12 postoperative hours.
Time Frame: Postoperative nausea and vomiting during the first 12 postoperative hours.
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine | 0.9% Sodium-chloride
Number analyzed (Participants) | 20 | 20
Participants | 16 | 19

ADVERSE EVENTS:
Time Frame: Intraop and 24 hours post-surgery.
Description: Record of vital signs was written in the anesthesia sheet.
  Non-serious adverse events were presented as follow:
  Hypotension Bradycardia Hypotension associated with bradycardia
Groups:
- Dexmedetomidine: After anesthesia induction, patients who were randomized to the Dexmedetomidine group, received a bolus of 1ug/kg in 10 minutes, followed by an infusion of 0.5ug/kg/h until the end of surgery. In the case of intraoperative increment of the blood pressure and/or heart rate more than 25% from its baseline, fentanyl 1ug/kg was administered.
  Dexmedetomidine: A bolus of 1ug/kg in 10 minutes, followed by an infusion of 0.5ug/kg/h until the end of surgery.
  Fentanyl: Intraoperative fentanyl was given in case of 25% increment in the blood pressure and/or heart rate in comparison to baseline (previous anesthesia induction).
  Morphine Sulfate: Boluses of 3mg of intravenous morphine were given in the postoperative acute care unit. Once the pain score was equal or less than 3/10 a patient-controlled analgesia pumps were installed and the patients were discharged to their room.
- 0.9% Sodium-chloride: After anesthesia induction, patients who were randomized to the Placebo group received a bolus and infusion of 0.9% normal saline at the same rate as the Dexmedetomidine group until the end of surgery. In the case of intraoperative increment of the blood pressure and/or heart rate more than 25% from its baseline, fentanyl 1ug/kg was administered.
  0.9% Sodium-chloride: The same dose used in the dexmedetomidine group (bolus and infusion).
  Fentanyl: Intraoperative fentanyl was given in case of 25% increment in the blood pressure and/or heart rate in comparison to baseline (previous anesthesia induction).
  Morphine Sulfate: Boluses of 3mg of intravenous morphine were given in the postoperative acute care unit. Once the pain score was equal or less than 3/10 a patient-controlled analgesia pumps were installed and the patients were discharged to their room.
Arm/Group | Dexmedetomidine | 0.9% Sodium-chloride
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 17/20 | 10/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexmedetomidine (N=20) | 0.9% Sodium-chloride (N=20)
Isolated hypotension (Cardiac disorders) | 2 (2) | 4 (4) — Isolated hypotension
Isolated Bradycardia (Cardiac disorders) | 7 (7) | 4 (4) — Isolated bradycardia
Hypotension associated with bradycardia (Cardiac disorders) | 10 (10) | 2 (2) — Hypotension and bradycardia combined

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes